CLINICAL TRIAL: NCT02606279
Title: Angiotensin Receptors and Age Related Mitochondrial Decline in HIV Patients
Acronym: RAS-HIV
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in study design and inability to recruit participants
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: WFUHS-28769
Record Dates: First submitted 2015-08-31; First posted 2015-11-17 (Estimated); Results first posted 2017-12-05 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-07

CONDITIONS: HIV; Aging; Sarcopenia; Angiotensin Receptor Antagonists
MeSH Terms: conditions — Sarcopenia | interventions — Valsartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo control (Placebo Comparator): 20 HIV-infected participants will be randomized into a blinded arm where they will receive 24 weeks of placebo therapy. During this time, they will undergo the same study procedures as the intervention arm.
  Interventions: Other: Placebo
- Valsartan (Experimental): 20 HIV-infected participants will be randomized into a blinded arm where they receive 24 weeks of valsartan therapy. For those subjects randomized to the valsartan group, they will receive valsartan 40 mg by mouth daily for 2 weeks, then increase to 80 mg by mouth daily for the remaining 22 weeks. During this time, they will undergo the same study procedures as the placebo arm.
  Interventions: Drug: valsartan

INTERVENTIONS:
Drug: valsartan — Valsartan will be given in increasing doses (from 40 mg to 80 mg) to those in the valsartan arm.
  Other Names: Diovan
  Arms: Valsartan
Other: Placebo
  Arms: Placebo control

SUMMARY:
This study is designed to evaluate specific factors in mitochondria that may precipitate premature aging and physical weakness in HIV patients. Angiotensin receptors 1 and 2 (AT1R and AT2R) are found in virtually every cell type. This study will evaluate how the relationships among these receptors in immune and skeletal muscle cells change with HIV, and how these changes might trigger mitochondrial dysfunction, declines in muscle strength, and cellular decline in people living with HIV.

DETAILED DESCRIPTION:
HIV related premature cellular aging and declines in mitochondrial function are closely linked. Dysfunctional mitochondria generate higher levels of reactive oxygen species (ROS) and provide less ATP supply cellular energy. Impaired turnover of damaged mitochondria leads to gradual but progressive decline in energy metabolism, increases in muscle fibrosis and clinically apparent weakness. The Renin Angiotensin System (RAS) is a central hormonal system that contributes to mitochondrial dysfunction and impacts both lifespan and function across multiple organ systems. Deletion of the angiotensin type 1 receptor (AT1R) results in a 25-30% extension of lifespan in mouse models, partly through increasing mitochondrial numbers. Blocking of AT1R reduces a number of age-related morbidities in mice, and in human studies. A plethora of data implicates RAS modulation in marked effects on fitness, frailty and beneficial responses to exercise in older adults. Despite this, there are virtually no data examining RAS biology in HIV+ vs. age-matched HIVsubjects, no data of RAS in relation to key HIV-specific variables (duration of HIV, treatment history, immune markers), and no data examining the effects of blocking AT1R on physical function in HIV infected subjects. In this study, we will examine the RAS and its contribution to premature mitochondrial failure in HIV patients. We will begin to fill this void by enrolling 40 HIV+ subjects in a randomized, double-blinded, placebo controlled pilot study of treatment with AT1R blocker to determine the feasibility of a larger trial, estimate effect size, assess the correlation of angiotensin receptor (AR) expression in peripheral blood cells and muscle cells, and the association of AR expression with physical function measures and immunity.

ELIGIBILITY:
Inclusion Criteria:

* able to provide informed consent
* able to attend an extended (~4 hour) Clinical Research Visit
* documented HIV seropositivity
* on a stable anti-retroviral therapy (ART) regimen for at least 12 months
* HIV plasma viral load < 50 copies/ml for at least 6 months
* Systolic blood pressure >110

Exclusion Criteria:

* creatinine > 1.5 ULN (or creatinine clearance < 60 ml/min)
* anti-hypertensive therapy with ACE-I or AT1R-blockers
* inability to perform functional measures (e.g. non-ambulatory without assistance, requires a prosthesis)
* recent (within 30 days) acute illness requiring medical therapy or hospitalization
* immunosuppressive agents (e.g. > 20 mg/d x 2 or more weeks of prednisone or equivalent, chemotherapy) in the last 6 months
* cancer requiring treatment w/in 3 yrs (except for non-melanoma skin cancer)
* blood thinning medications such as Coumadin or Plavix or a bleeding disorder such as hemophilia that could cause complications during muscle biopsies
* pregnancy (will provide urine test for females of child bearing potential)
* regular use of non-steroidal anti-inflammatory drugs or other immune modulating agents.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2014-07; Primary Completion 2016-08-04 (Actual); Study Completion 2016-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine R Schafer, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Control: 20 HIV-infected participants will be randomized into a blinded arm where they will receive 24 weeks of placebo therapy. During this time, they will undergo the same study procedures as the intervention arm.
  Placebo
Period: Overall Study
Arm/Group | Placebo Control | Valsartan
Started | 0 | 1
Completed | 0 | 0
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Gender, Race, and Ethnicity info not released due to confidentiality issues in this small sample of n=1
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Control | Valsartan | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 1 | 1
  >=65 years |  | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male |  | 0 | 0
  Female |  | 0 | 0
  Prefers not to identify |  | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 0 | 0
  Not Hispanic or Latino |  | 0 | 0
  Unknown or Not Reported |  | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 0 | 0
  White |  | 0 | 0
  More than one race |  | 0 | 0
  Unknown or Not Reported |  | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 400m Walk
Description: Measured by time to finish 400 meter walk
Time Frame: 3, 6, and 9 months post-enrollment
Population: Participant did not complete visits, data not collected.
Arm/Group | Placebo Control | Valsartan
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Change From Baseline in Grip Strength
Description: Measured by dynamometer measurement of grip strength
Time Frame: 3, 6, and 9 months post-enrollment
Population: Participant did not complete visits, data not collected.
Arm/Group | Placebo Control | Valsartan
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Change From Baseline in Quantity of AT1R and AT2R on Monocytes
Description: Measured by using qPCR and western blot. (Units are arbitrary units)
Time Frame: 3, 6, and 9 months post-enrollment
Population: Participant did not complete visits, data not collected.
Arm/Group | Placebo Control | Valsartan
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change From Baseline in Frailty Status
Description: Evaluated by measurements of grip strength, walking speed and questionnaires
Time Frame: 3, 6, and 9 months post-enrollment
Population: Participant did not complete visits, data not collected.
Arm/Group | Placebo Control | Valsartan
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Placebo Control | Valsartan
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No